CLINICAL TRIAL: NCT02566863
Title: Haemodynamic Effect of Dexmedetomidine in Relation to Autonomic System Activity
Brief Title: Haemodynamic Effect of Dexmedetomidine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Magdalena Wujtewicz, M.D., Ph.D, Medical University of Gdansk
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GUMed-Wu-003
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Haemodynamic Effects of Dexmedetomidine
Keywords: dexmedetomidine; heart rate; heart rate variability
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexmedetomidine (Experimental): Dexmedetomidine, 1 mcg/kg over 10 minutes, followed by a maintenance infusion, given to achieve sedation for eye surgery procedure
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — 1 mcg/kg over 10 minutes, followed by a maintenance infusion titrated to achieve desired clinical effect - Richmond Agitation Scale between 0 and (-) 3. Holter ECG recording before start of infusion and during infusion for 25 minutes.
  Other Names: Dexdor; Precedex

SUMMARY:
Dexmedetomidine, selective alfa2 receptors agonist produces sympatholysis. As a result heart rate decreases. With low doses blood pressure also decreases, with higher dosing - systematic vascular resistance increases. The indication for the drug is to produce sedation during surgical procedures and in ICU patients.

The aim of a study is to verify, whether the haemodynamic effect (heart rate, blood pressure and heart rate variability during drug infusion) depend on pre-drug autonomic system activity. Autonomic system activity is assessed using heart rate variability (HRV)measurement before drug injection and during drug infusion. Heart rate and blood pressure measured before and during drug infusion will be analysed.

HRV measurement analysis will be based on continuous Holter ECG recording, taken before drug injection and during its infusion. 5 minutes intervals will be analysed , using Frequency Domain Measures of HRV. Surgical procedure will start after measurement have been taken.

ELIGIBILITY:
Inclusion Criteria:

* patients classified with American Society of Anesthesiologists Physical Status Classification System as 1 or 2 status
* planned eye surgery under sedation

Exclusion Criteria:

* patient's refusal
* contraindications to dexmedetomidine
* diseases/drugs that influence on autonomic nervous system activity

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-06; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Changes of haemodynamics and heart rate variability parameters | up to 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena A Wujtewicz, M.D, Principal Investigator — Department of Ophthalmology, Medical University of Gdańsk
Locations (1):
- Medical University of Gdansk, Gdansk, Poland